CLINICAL TRIAL: NCT04651413
Title: Can Quantitative (Real-time) Polymerase Chain Reaction (PCR) Cycle Threshold (Ct) Values be Used to Predict Poor Outcomes for Patients Infected With SARS-CoV-2? A Local Exploratory Sub-study at The University Hospitals of North Midlands NHS Trust in Collaboration With the International Severe Acute Respiratory and Emerging Infection Consortium (ISARIC) COVID-19 Trial
Brief Title: PCR Cycle Threshold Values and COVID-19 Outcomes
Status: Completed | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 286389
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2020-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 Ct Value: All patients enrolled onto the ISARIC COVID-19 trial at The University Hospitals of North Midlands NHS Trust between the period 1st February 2020 to 1st July 2020 will be included in this study, provided that a laboratory cycle threshold (Ct) value is available.
  Interventions: Diagnostic Test: PCR Value

INTERVENTIONS:
Diagnostic Test: PCR Value — Data collection and interpretation

SUMMARY:
This is a retrospective observational study. The study will use high quality, reliable data that has already been collected for the ISARIC 4C COVID-19 study in order to analyse the relation between predictor variables (laboratory polymerase chain reaction [PCR] cycle threshold [Ct] values) and outcomes for COVID-19 disease within a hospitalised population.

DETAILED DESCRIPTION:
Currently, in the United Kingdom, the recommended method for diagnostic testing and screening for COVID-19 is quantitative (real-time) reverse transcription polymerase chain reaction (PCR) analysis of viral RNA extracted from upper respiratory tract samples. A positive result indicates that SARS-CoV-2 RNA has been detected with a cycle threshold (Ct) value of less than 38 cycles of amplification (n.b. this is a locally agreed value, which is based on analysis of proficiency testing performance and other local testing data. Cycle threshold (Ct) values inversely correlate to the amount of target nucleic acid in the sample. Thus, a lower cycle threshold (Ct) value indicates a greater amount of target nucleic acid in a sample i.e. a higher viral load.

A recent scoping literature review has revealed only a handful of published studies to date that explore an association between cycle threshold (Ct) values and disease severity or clinical outcome in patients infected with the SARS-CoV-2 virus. The majority of these studies have been conducted in China with small patient sample sizes. Thus, a larger-scale study which explores the relationship between viral load and disease severity is required; indeed, the World Health Organization (WHO) has recently highlighted this as an area which needs further research.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (aged 18 years and over) patients presenting to UHNM with confirmed SARS-CoV-2 infection AND who are enrolled onto the ISARIC COVID-19 study.
2. Patients who have undergone an initial diagnostic or screening test for SARS-CoV-2 (from an upper respiratory tract sample) AND a cycle threshold (Ct) value is available on the UHNM laboratory database.

Exclusion Criteria:

1. Paediatric patients (under 18 years).
2. Patients without a PCR Ct result on the UHNM laboratory database
3. Patients without confirmed SARS-CoV-2 infection
4. Patients who were not enrolled in to the ISARIC COVID-19 study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults (aged 18 years and over) patients presenting to UHNM with confirmed SARS-CoV-2 infection and who are enrolled onto the ISARIC 4C COVID-19 study. These patients must also have undergone an initial diagnostic or screening test for SARS-CoV-2 (from an upper respiratory tract sample) and a cycle threshold (Ct) value is available on the UHNM laboratory database.
Sampling Method: Probability Sample
Enrollment: 934 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Determine if there is an inverse correlation with risk of poor outcome including admission to intensive care; mechanical ventilation and 28-day mortality. | 01/02/2020 to 01/07/2020
  Determine if cycle threshold (Ct) levels are an independent predictor for:
  I. Hypoxia resulting in oxygen dependency or oxygen saturations < 92%, at admission and at any other point during the episode of care; II. admission to intensive care; III. mechanical ventilation and

SECONDARY OUTCOMES:
Differences in cycle threshold (Ct) levels amongst patients with community acquired SARS-CoV-2 | 01/02/2020 to 01/07/2020
  Determine if sociodemographic factors are significantly associated with lower cycle threshold (Ct) levels.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kemp, Principal Investigator — UHNM
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No